CLINICAL TRIAL: NCT01800513
Title: EVAULATION OF IMPLANTATION AND PREGNANCY AFTER ENDOMETRIAL INJURY VIA ENDOMETRIAL PIPELLE BIOPSY IN THE CYCLE PRIOR TO IVF: A RANDOMIZED, SINGLE-BLINDED, CONTROLLED TRIAL.
Brief Title: Endometrial Biopsy Prior to IVF in Those Patients With Prior Implantation Failure
Acronym: EMBX/IVF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shady Grove Fertility Reproductive Science Center (Other)
Responsible Party: Principal Investigator, Ryan Heitmann, REI Clinical Fellow, Shady Grove Fertility Reproductive Science Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SGFRSC EMBX 2013
Record Dates: First submitted 2013-02-21; First posted 2013-02-27 (Estimated); Last update posted 2013-02-27 (Estimated); Status verified 2013-02

CONDITIONS: Implantation Failure; Infertility
Keywords: Implantation Failure; In-vitro Fertilization; Infertility; Endometrial Biopsy
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Endometrial Biopsy (Experimental): Subjects will have a vaginal speculum placed and visualization of the cervix will be obtained. The cervix will be cleaned with betadine (or hibiclens for those with an iodine allergy). Those randomized to the treatment arm (endometrial biopsy) will have an endometrial pipelle (Endocell, Wallach, Orange, Connecticut) inserted gently through the cervix into the uterus. Two passes will be performed with the pipelle catheter. For each pass the catheter will be rotated and scraped 4 times, once in each quadrant.
  Interventions: Procedure: Endometrial Biopsy
- Control (Sham Comparator): Those randomized to the control group will have a small cotton swab placed gently into the cervix. No tissue will be obtained with this method. The randomization to a placebo control is necessary to prove that any positive effects seen are due to the biopsy and not just random chance.
  Interventions: Procedure: Sham Procedure

INTERVENTIONS:
Procedure: Endometrial Biopsy
  Other Names: Endometrial Pippelle Biopsy Catheter
  Arms: Endometrial Biopsy
Procedure: Sham Procedure
  Arms: Control

SUMMARY:
This proposed research is a single center, prospective, single-blinded, randomized controlled trial, designed to evaluate IVF pregnancy outcomes following endometrial injury in 254 patients with implantation failure. Patients will be identified during their work-up and treatment at Shady Grove Fertility Reproductive Science Center. Only Shady Grove patients are eligible for the study. The investigators hypothesize in patients with one or more previous failed day 5 blastocyst transfers, injury to the endometrium via endometrial biopsy will improve clinical pregnancy outcomes compared to controls.

DETAILED DESCRIPTION:
Despite advances in assisted reproductive technologies; implantation failure in patients undergoing in-vitro fertilization (IVF) is frequent. Unfortunately, few treatments exist except for the use of a gestational carrier. There have been a number of recent clinical studies demonstrating that local injury to the endometrium results in improved clinical pregnancy outcomes for patients with a history of implantation failure. However, not all studies have shown a beneficial effect, and those demonstrating benefit have been limited by small sample sizes, and considerable heterogeneity in the procedures and populations evaluated. A recent meta-analysis synthesized the available data concluded that a large, prospective, well-designed randomized trial is desperately needed to definitively assess this new possible treatment. If these preliminary findings from previous trials are confirmed, this practice could be applied in the clinical setting to help patients suffering from repeated implantation failures.

ELIGIBILITY:
Inclusion Criteria:

* Women age 18-37
* One or more previous implantation failures with autologous fresh or frozen blastocyst transfer
* Undergoing fresh autologous IVF cycle
* No other current uterine (i.e.: uterine fibroids, polyps), hematologic, or genetic causes for infertility and implantation failure
* One or more good quality blastocyst(s) available for transfer

Exclusion Criteria:

* Those unable to comprehend the investigational nature of the proposed study
* Positive pregnancy test
* Possible causes for impaired implantation (systemic disease, endometriosis, ultrasound evidence of current hydrosalpinx, uterine polyps, uterine myomas (fibroids), uterine cavity malformations or Asherman's syndrome)
* Poor responders, defined as FSH >12 on day 3 or less than 4 follicles on a previous IVF cycle
* BMI >30 or <18

Ages: 18 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 254 (Estimated)
Dates: Start 2013-02; Primary Completion 2014-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
The primary outcome measurement in this study is clinical pregnancy rate, which is defined as identification of a fetal heart beat on ultrasound. | 8-10 weeks after embryo transfer

SECONDARY OUTCOMES:
implantation rate | 8-10 weeks after embryo transfer
miscarriage rate | 2 years
multiple gestation rate | at delivery
endometrial thickness during stimulation | during stimulation
Live Birth rate | 10 months after IVF cycle

CONTACTS AND LOCATIONS:
Overall Officials: Erin F Wolff, M.D., Principal Investigator — Shady Grove Fertility
Locations (1):
- Shady Grove Fertility Reproductive Science Center, Rockville, Maryland, United States

REFERENCES:
- See also: Shady Grove Fertility Home Page — http://www.shadygrovefertility.com